CLINICAL TRIAL: NCT05993390
Title: Effect of Neuromuscular Reversal Agents on Time for Neurological Assessment After Endotracheal Intubation in Critically Ill Patients
Brief Title: Pharmacological Reversal of Neuromuscular Blockade in Critically Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-2306-197-1445
Record Dates: First submitted 2023-07-19; First posted 2023-08-15 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Neuromuscular Blockade; Critical Illness; Neurologic Findings
Keywords: Reversal of neuromuscular blockade; Neurologic assessment; Endotracheal intubation; Critically ill patient
MeSH Terms: conditions — Critical Illness; Neurologic Manifestations | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sugammadex group (Experimental): Patient is intubated with etomidate 0.1~0.2mg/kg and rocuronium 1mg/kg. 30 minutes after rocuronium administration, patient is administered sugammadex 1mg/kg. Glasgow coma scale as neurologic assessment is assessed at 10-minute intervals before intubation, and at 5-minute intervals up to 30 minutes after administration of sugammadex. After 30 minutes, the assessments are conducted at 10-minute intervals. Additionally, if the patient spontaneously opens their eyes, the GCS is assessed at that specific moment. The GCS evaluation continues until the patient reaches a point of responsiveness, indicated by a Motor score of 6 on the GCS.
  Interventions: Drug: Sugammadex
- Neostigmine group (Experimental): Patient is intubated with etomidate 0.1~0.2mg/kg and rocuronium 1mg/kg. 30 minutes after rocuronium administration, patient is administered neostigmine 0.05mg/kg + glycopyrrolate 0.01mg/kg. Glasgow coma scale as neurologic assessment is assessed at 10-minute intervals before intubation, and at 5-minute intervals up to 30 minutes after administration of neostigmine. After 30 minutes, the assessments are conducted at 10-minute intervals. Additionally, if the patient spontaneously opens their eyes, the GCS is assessed at that specific moment. The GCS evaluation continues until the patient reaches a point of responsiveness, indicated by a Motor score of 6 on the GCS.
  Interventions: Drug: Neostigmine
- Control group (No Intervention): Patient is intubated with etomidate 0.1~0.2mg/kg and rocuronium 1mg/kg. Glasgow coma scale as neurologic assessment is assessed at 10-minute intervals before intubation, and at 5-minute intervals up to 60 minutes after intubation. After 60 minutes, the assessments are conducted at 10-minute intervals. Additionally, if the patient spontaneously opens their eyes, the GCS is assessed at that specific moment. The GCS evaluation continues until the patient reaches a point of responsiveness, indicated by a Motor score of 6 on the GCS.

INTERVENTIONS:
Drug: Sugammadex — Intravenous administration of sugammadex 2mg/kg.
  Arms: Sugammadex group
Drug: Neostigmine — Intravenous administration of neostigmine 0.05mg/kg with glycopyrrolate 0.01mg/kg
  Arms: Neostigmine group

SUMMARY:
The goal of this clinical trial is to compare the effect of use of reversal agents for neuromuscular blockade in critically ill patients on time for neurological assessment after endotracheal intubation

The main questions it aims to answer are:

* The use of reversal agents for neuromuscular blockade after endotracheal intubation may reduce the time for neurological assessment.
* The types of reversal agents for neuromuscular blockade may affect the time for neurological assessment.

Participants will receive different reversal agents or no medications based on the assigned groups. Thirty minutes after intubation using rocuronium, medication is administered, and the time of initial confirmation of eye opening and movement is recorded.

Researchers will compare 3 groups (sugammadex, neostigmine and control(no medication) to see the difference of time for neurological assessment after endotracheal intubation.

DETAILED DESCRIPTION:
Patients who agree to participate in the study will be randomized to the sugammadex group, neostigmine group, or control group.

Randomization will be performed by an independent investigator. Patient, medical staff performing patient evaluation are masked for the assignment otherwise the medical staff administering medications to patient is not blinded.

An independent investigator, who is not included in this study, will provide the assignment result to the medical staff administering medications to patient.

1. Neurologic assessment

   The point at which first available neurologic assessment is defined as the point at which the patient is able to move on command (Motor score of 6 on the GCS), and the GCS will be assessed until that point.

   Regardless of randomization outcome, all patients will be monitored for GCS and monitored for processed EEG and cerebral regional oxygen saturation prior to intubation.

   Assessment of GCS before administration of sedatives for endotracheal intubation, every 10 minutes after intubation, before administration of study medications, every 5 minutes until 30 minutes after administration of study medications, and every 10 minutes after 30 minutes, with additional assessments at that time if spontaneous eye opening occurs. The GCS will be assessed until directed movement is possible (Motor score of 6 on the GCS).

   Eye opening response: If there is no response after 2 repetitions of 'OOO, please open your eyes', the response is evaluated with 2 repetitions of the stimulus of pressing the thumb nail. If the subject opens his/her eyes spontaneously, skip this assessment.

   Motor response: 'Please make a fist' and 'Please open your fist' are performed twice, and if there is no response, the stimulus of pressing the thumb nail is performed twice to assess the response.
2. Processed EEG and cerebral regional oxygen saturation

   Processed EEG using Masimo's Next Generation SedLine® Brain Function Monitoring, and cerebral regional oxygen saturation using Masimo's O3® Regional Oximetry is monitored and recorded.

   Processed EEG and cerebral regional oxygen saturation will be recorded at 10 minute intervals from before sedation for intubation until neurological function can be assessed.
3. Neuromuscular function monitoring

   Utilized by the Philips Intellivue NMT(neuromuscular transmission) monitor. Monitor every 5 minutes beginning 30 minutes after Rocuronium dosing and discontinue monitoring if eyes open spontaneously (Eye score of 4 on GCS).
4. Endotracheal intubation 100% oxygen is delivered via a facial fitting mask. Patients who have been maintained on oxygen via a high-flow nasal cannula are given 100% oxygen with a flow rate of 60 L/min.

   Sedation is administered with etomidate 0.1-0.2 mg/kg, and endotracheal intubation is performed with rocuronium 1 mg/kg once the patient's loss of consciousness is confirmed.
5. Drug Administration

   Sugammadex treatment group

   Neuromuscular function monitoring is performed every 5 minutes starting 30 minutes after rocuronium administration.

   Sugammadex 0.2 mg/kg 30 minutes after rocuronium is administered, after GCS assessment and neuromuscular function monitoring.

   Processed EEG and cerebral regional oxygen saturation levels at the time of sugammadex administration is recorded.

   Neostigmine group Neuromuscular function monitoring is performed every 5 minutes starting 30 minutes after rocuronium administration.

   Administer neostigmine 0.05 mg/kg + glycopyrrolate 0.01 mg/kg after rocuronium is administered, after GCS assessment and neuromuscular function monitoring.

   Processed EEG and cerebral regional oxygen saturation levels at the time of sugammadex administration is recorded.

   Control group Processed EEG and cerebral regional oxygen saturation levels at the time of sugammadex administration is recorded.
6. GCS assessment and neuromuscular function monitoring is performed 30 minutes after rocuronium administration, and processed EEG and cerebral regional oxygen saturation levels is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 19 years of age or older who were intubated after admission to the intensive care unit.

Exclusion Criteria:

* Patients younger than 19 years of age
* Patients who are not neurologically evaluable or have concomitant neurologic dysfunction
* Patients with neuromuscular disorder
* Patients with a history of drug allergic reactions to sugammadex or neostigmine
* Patients taking or planning to take toremifene, fusidic acid, or hormonal contraceptives

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Time from administration of neuromuscular blocker to the first available neurologic assessment (in minutes) | Time from administration of neuromuscular blocker to first available neurologic assessment (Motor score 6 on GCS, in minutes), assessed up to 48 hours.
  Time from administration of neuromuscular blocker to the first time the patient is able to make a directed movement (Motor score 6 on GCS), assessed up to 48 hours.

SECONDARY OUTCOMES:
Time from administration of neuromuscular blocker to first available spontaneous eye opening (in minutes) | Time from administration of neuromuscular blocker to first time the patient is able to open eyes spontaneously (Eye score 4 on GCS, in minutes), assessed up to 48 hours.
  Time from administration of neuromuscular blocker to first time the patient is able to open eyes spontaneously (Eye score 4 on GCS), assessed up to 48 hours.
Changes of Patient State index (PSi) values | Before intubation (Time 0), Time 10/20/30/35/40/45/50/55/60/70/80/90 minutes
  Changes of Patient State index (PSi) values
Changes of regional cerebral oxygen saturation (O3) values | Before intubation (Time 0), Time 10/20/30/35/40/45/50/55/60/70/80/90 minutes
  Changes of regional cerebral oxygen saturation (O3) values
Time from intubation to extubation | Date of the patient extubated, up to 1 month
  Time from intubation to extubation, up to 1 month
Total length of hospital stay | Date of discharge from the hospital, up to 1 month
  Total length of hospital stay, up to 1 month
Total length of intensive care unit(ICU) stay | Date of discharge from the ICU, up to 1 month
  Total length of intensive care unit(ICU) stay, up to 1 month
In-ICU mortality | Date of death from any cause in ICU, up to 1 month
  In-ICU mortality, up to 1 month
In-hospital mortality | Date of death from any cause in hospital, up to 1 month
  In-hospital mortality, up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ho Geol Ryu, M.D., Ph.D, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No